CLINICAL TRIAL: NCT01457391
Title: A Stage II Efficacy Study of Cognitive Behavioral Therapy for PTSD in Community Addiction Treatment
Brief Title: Cognitive Behavioral Therapy (CBT) for Posttraumatic Stress Disorder (PTSD) in Community Addiction Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Mark McGovern, Professor of Psychiatry and of Community and Family Medicine, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5R01DA027650 (NIH); 5R01DA027650 (NIH)
Record Dates: First submitted 2011-10-04; First posted 2011-10-24 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Stress Disorders, Post-Traumatic; Substance-Related Disorders
Keywords: cognitive behavioral therapy; addiction; posttraumatic stress disorder (PTSD)
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Substance-Related Disorders; Behavior, Addictive | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cognitive Behavioral Therapy (Experimental): Cognitive Behavioral Therapy (CBT) is a non-exposure based manual-guided individual therapy. CBT for PTSD consists of 3 learning and skill components designed to improve PTSD symptoms and substance use: 1) Patient education about PTSD and its relation to substance use and treatment; 2) Breathing retraining: A behavioral anxiety reduction skill; and 3) Cognitive restructuring: A cognitive approach and functional analysis of the link among emotions, cognitions and situations.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Individual Addiction Counseling (Active Comparator): Individual Addiction Counseling (IAC) was adapted from the Individual Drug Counseling (IDC) manual used in the NIDA Cocaine Collaborative Study. IAC is a manual-guided treatment that focuses on substance use and history of use, consequences of use and denial, developing strategies for relapse prevention, and facilitation of connection with peer recovery support groups, specifically twelve step groups. The current adaptation of IAC modified the IDC manual by broadening the focus to include drugs other than cocaine, as well as alcohol.
  Interventions: Behavioral: Individual Addiction Counseling
- Treatment-as-usual (Active Comparator): Treatment-as-usual (TAU) is the typical intensive outpatient (IOP) treatment that the patient would receive ordinarily at the identified addiction treatment program. Each TAU service operates using the American Society of Addiction Medicine criteria for Level II Intensive Outpatient services: 9-12 hours per week; group and individual sessions focused on motivation to address substance use, education about the consequences of substance use on major life areas, education about the disease concept and brain changes associated with addiction, exposure to information about social and family relationships and recovery, and relapse prevention skills.
  Interventions: Behavioral: Treatment-as-usual

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Individual CBT, approx. 12 sessions, one session per week
  Other Names: CBT for PTSD; Integrated Cognitive Behavioral Therapy; ICBT; CBT
  Arms: Cognitive Behavioral Therapy
Behavioral: Individual Addiction Counseling — Individual therapy, approx. 12 sessions, one session per week
  Other Names: IAC
  Arms: Individual Addiction Counseling
Behavioral: Treatment-as-usual — Individual or group therapy, approx. 9-12 hours per week, multiple times a week for 2 months
  Other Names: TAU
  Arms: Treatment-as-usual

SUMMARY:
The purpose of this phase of the study is to assess the efficacy of CBT for PTSD, as delivered by routine addiction counselors in community treatment programs, and to compare CBT for PTSD with both Individual Addiction Counseling (IAC) and Treatment as Usual (TAU) on the primary outcomes.

DETAILED DESCRIPTION:
The main hypothesis being tested is that a cognitive behavioral therapy (CBT) for posttraumatic stress disorder (PTSD) can improve treatment retention and outcomes for both posttraumatic stress and substance use disorders. The investigators have completed the Stage I Safety & Practicality Study, Feasibility Study and Pilot Randomized Controlled Study (comparing CBT for PTSD to versus a control condition) and for all studies found that CBT for PTSD was safe and effective in reducing PTSD symptoms, improving retention, and in reducing substance use. The present study proposes to continue testing the hypotheses by evaluating and comparing the PTSD, retention and substance use outcomes resulting from CBT versus a control condition and to treatment as usual. This is termed a "Stage II Efficacy Study" of behavioral therapy development and requires comparing the investigational treatment (CBT) with a control treatment, within the context of addiction treatment-as-usual (intensive outpatient programs). This is a larger randomized controlled trial in response to the outcomes of the pilot trial. The proposed research will evaluate the efficacy of a relatively simple, manual-guided cognitive behavioral therapy (CBT) for PTSD. CBT for PTSD has been designed and developed for delivery by counselors employed in community addiction treatment programs and offered in conjunction with standard community addiction treatment. Outpatients at each of 7 community addiction treatment programs, diagnosed with current PTSD will be randomly assigned to receive either: 1) CBT for PTSD in conjunction with standard treatment-as-usual (TAU) (n=76); 2) A manual-guided individual addiction counseling (IAC) adapted from the Individual Drug Counseling Manual in conjunction with TAU (n=76); or 3) TAU (n=76) without additional individual treatment for either PTSD or substance use disorders. Treatment will be delivered by frontline counselors from and onsite in the addiction treatment programs.

Our objective is to test the following specific hypotheses:

1. Patients exposed to CBT for PTSD plus treatment-as-usual (TAU) will show significantly greater improvements in PTSD symptom severity relative to patients in the other two interventions (IAC+TAU and TAU alone) at both the three-month and six-month follow-ups. The IAC+TAU condition will show no greater reduction in PTSD symptom severity than the TAU condition at both the three-month and six-month follow-ups.
2. Patients receiving the CBT for PTSD plus TAU will manifest equivalent reductions in substance use severity (drug and/or alcohol) to patients in the IAC+TAU intervention conditions at both the three-month and six-month follow-ups. CBT and IAC are both active treatments targeting substance use symptoms. The CBT+TAU and IAC+TAU condition patients will exhibit greater reductions in substance use than patients in the TAU condition at both the three-month and six-month follow-ups.
3. Patients in the CBT condition will have better retention in the addiction treatment program relative to the IAC+TAU and TAU alone intervention conditions. IAC+TAU will have better retention in the addiction treatment program than TAU alone.

This study involves a three-group repeated measure design. Within the NIDA stage model, it is a randomized controlled trial with a matched-attention control condition. The investigators plan to examine the outcomes associated with the intervention versus control condition versus treatment-as-usual among patients receiving outpatient addiction treatment services (intensive outpatient programs). The investigators will employ assessments at baseline, three-month follow-up, and six-month follow-up. Eligible subjects will be randomly assigned to the study CBT therapy (plus addiction treatment-as-usual), the matched attention control condition (individual addiction counseling [IAC] plus addiction treatment-as-usual) or the addiction treatment-as-usual, and all will be followed for the research assessments regardless of whether they drop out of treatment early (whenever possible).

Patients admitted to the participating addiction treatment programs are routinely screened for PTSD using a brief self-report survey, the PTSD checklist (PCL). These forms are collected by clinical staff of teh treatment program and scored for PTSD diagnostic criteria. Patients scoring 44 or greater on the PCL are approached by a clinic staff about potential interest in the study. If they wish to learn more about the study, research coordinator (or on-site employee) is contacted, a suitable time arranged, and the patient engaged in the process of informed consent.

If consent is granted, the subjects completes the baseline assessment. The baseline assessment consists of measures gathered via interview by a member of the research team, self-administered surveys completed directly by the subject, and review of the subject's medical record to extract demographic, substance use, and treatment history information, as well as chart diagnoses.

The interview portion of the assessment consists of:

* Standardized interviews designed to assess PTSD and other commonly associated axis I DSM-IV diagnoses: Clinician Administered PTSD Scale (CAPS) and the Structured Clinical Interview for DSM-IV (SCID).
* A urine screen and breathalyzer to test for alcohol and other drugs.
* Standardized follow-back method for gathering data on recent alcohol and drug use: Time-line Follow-back Calendar (TLFB).

The self-administered portion of the assessment consists of measures designed to assess:

* Alcohol and drug use, as well as associated problems in other life areas such as medical, employment, legal, social, and psychiatric: Addiction Severity Index (ASI)
* Treatment utilization: Recent Treatment Survey (RTS).

If the subject continues to meet criteria for PTDS (i.e. the CAPS interview confirms diagnosis of DSM-IV PTSD, with symptom severity at 44 or higher), he or she is randomized to receive the study CBT therapy, control condition (IAC), or treatment-as-usual (TAU).

Research assessments are then also conducted at three months and six months post baseline assessment. This follow-up assessments will consist of the same measures administered at baseline, with the exception of the SCID interview.

The investigators plan to randomize approximately 228 subjects in the study (76 to CBT, 76 to IAC, and 76 to TAU).

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old;
2. Actively enrolled in outpatient addiction services and meets criteria for substance use disorder;
3. Screened positive for PTSD (results of PCL show a likely Criterion A Traumatic Event and a score equal to or greater than 44);
4. Willing and able to provide informed consent to participate in the study;
5. Diagnosis of PTSD verified by the CAPS and total symptom score equal to or greater than 44;

Exclusion Criteria:

1. Acute psychotic symptoms (however, persons with a psychotic disorder are eligible if their symptoms are stable and they are well connected with appropriate mental health services);
2. Psychiatric hospitalization or suicide attempt in the past month (however, if the hospitalization or attempt was directly related to substance intoxication or detoxification and the person is currently stable, they are eligible);
3. Medical and/or legal situations are unstable such that ability to participate in the full duration of the study seems unlikely.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 443 (Actual)
Dates: Start 2010-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Decrease from baseline in PTSD symptom severity (Clinician Administered PTSD Scale (CAPS) score (30 day)) at 3-months and at 6-months | Baseline, 3-month, & 6-month follow-ups
Decrease from baseline in positive toxicology screens (urine drug screen and breathalyzer) at 3-months and at 6-months | Baseline, 3-month, & 6-month follow-ups
Decrease from baseline in drug and alcohol symptom severity (Addiction Severity Index (ASI)-Self Administered (30 day)) at 3-months and at 6-months | Baseline, 3-month, & 6-month follow-ups
Decrease from baseline in frequency of substance use (Timeline Follow-Back (TLFB) Interview (90 day)) at 3-months and at 6-months | Baseline, 3-month, & 6-month follow-ups

SECONDARY OUTCOMES:
Difference in treatment retention (continuation and completion of ICBT or IAC) | From date of treatment commencement until treatment completion, assessed up to approx. 12 weeks
Therapist adherence and competence (ICBT or IAC) | Duration of study intervention

CONTACTS AND LOCATIONS:
Overall Officials: Mark P. McGovern, Ph.D., Principal Investigator — Geisel School of Medicine at Dartmouth College
Locations (4):
- United States (4):
  - Central Vermont Substance Abuse Services, Berlin Corners, Vermont
  - Brattleboro Retreat, Brattleboro, Vermont
  - Howard Center, Burlington, Vermont
  - Evergreen - Rutland Mental Health, Rutland, Vermont

REFERENCES:
- [Derived] Meier A, McGovern MP, Lambert-Harris C, McLeman B, Franklin A, Saunders EC, Xie H. Adherence and competence in two manual-guided therapies for co-occurring substance use and posttraumatic stress disorders: clinician factors and patient outcomes. Am J Drug Alcohol Abuse. 2015;41(6):527-34. doi: 10.3109/00952990.2015.1062894. Epub 2015 Aug 18. PMID 26286351
- [Derived] McGovern MP, Lambert-Harris C, Xie H, Meier A, McLeman B, Saunders E. A randomized controlled trial of treatments for co-occurring substance use disorders and post-traumatic stress disorder. Addiction. 2015 Jul;110(7):1194-204. doi: 10.1111/add.12943. PMID 25846251